CLINICAL TRIAL: NCT06172751
Title: TrinetX Study of Hypereosinophilic Syndrome (HES) Without an Identifiable Non-haematological Secondary Cause
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3254R00004
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Hypereosinophilic Syndrome (HES)
MeSH Terms: conditions — Hypereosinophilic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- anti-IL-5/IL-5R therapy: Patients initiated anti-IL-5/IL-5R therapy
  Interventions: Other: no intervention
- other therapies: Patients initiated other therapies.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — not applicable, this is an observational retrospective data analysis study; no interventions in the study
  Groups: anti-IL-5/IL-5R therapy
Other: no intervention — not applicable, this is an observational retrospective data analysis study; no interventions in the study
  Groups: other therapies

SUMMARY:
The purpose of this study is to build the knowledge base on clinical characteristics, clinical management, and treatment outcomes of HES.

DETAILED DESCRIPTION:
Retrospective database analysis using TriNetX database to describe HES patient characteristics, journey, and disease burden.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis record of HES (ICD-10-CM D72.11) anytime during 01 October 2020 to 30 June 2023
* At least 12 months of patient insurance record prior to first HES record.

Exclusion Criteria:

* Any mutation in PDGFRA, PDGFRB or FGFR1 genes (to exclude clonal HES).
* History of BCR-ABL tyrosine kinase inhibitor use: imatinib, dasatinib, nolitinib, bosutinib, ponatinib, asciminib (to exclude clonal HES)
* History of myeloid leukemia, myeloproliferative disorder, myelodysplastic disorder, myelomonocytic leukemia, acute erythroid leukemia, acute megakaryoblastic leukaemia, acute panmyelosis with myelofibrosis, and other specified leukaemias (to exclude reactive HES)
* History of helminthiasis or use of anthelmintic medication (to exclude reactive HES)
* History of autoimmune disease (to exclude reactive HES)
* History of use of specific drugs: antiepileptics, sulfonamides, allopurinol, and immune checkpoint inhibitors (to exclude reactive HES)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is patients with HES during the period 01 October 2020 to 30 June 2023 available in TrinetX database (US).
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Comorbidities prior to first HES record | 01 October 2020- the most recent data available in 2023
  To describe clinical characteristics of patients with HES.
Other eosinophilic conditions | 01 October 2020- the most recent data available in 2023
  To describe the clinical characteristics of HES patients.
Organ system with HES signs and/or symptoms | 01 October 2020- the most recent data available in 2023
  To describe the disease burden of HES.
Number of organ systems with HES signs and/or symptoms | 01 October 2020 - the most recent data available in 2023
  To describe the disease burden of HES.

SECONDARY OUTCOMES:
Demographic characteristics | 01 October 2020- the most recent data available in 2023
  To describe the demographic characteristics of HES patients and sub-group analysis patients.
Patient journey in diagnostic phase | 01 October 2020 - the most recent data available in 2023
  To describe the patient journey in diagnostic phase and in sub-group analysis.
HES and non-HES therapies & treatment pattern | 01 October 2020 - the most recent data available in 2023
  To describe the treatment pattern of HES patients and sub-group analysis patients.
Clinical outcomes | 01 October 2020 - the most recent data available in 2023
  To describe clinical outcome pre and post index date and compare between biologics and patients treated with anti-IL-5/IL-5Rα therapies.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Cambridge, Massachusetts, United States

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3254R00004&attachmentIdentifier=937528c6-d4bf-4827-9f4c-53e440c1668c&fileName=D3254R00004_AZ_TriNetX_HES_study_report_synopsis_redacted.pdf&versionIdentifier=